CLINICAL TRIAL: NCT01837524
Title: The KP Personal Shopper: A Pilot to Improve the Impact of Dietary Advice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00003988
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2014-01

CONDITIONS: Overweight; Obesity
Keywords: Dietary advice; Nutritional knowledge; Self-efficacy; Nutrition
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grocery-Store-Based Visit Arm (Experimental): 25 participants will be randomized to this arm. They will receive a baseline 30-minute phone call with the study dietitian to determine their current health problems, dietary patterns, shopping and cooking habits and health goals. They will then have 3 in-person visits with the dietitian conducted during grocery shopping trips at a local supermarket. These in-person visits will be conducted monthly over a 3 month period. The information delivered in the visits will be similar in content to that delivered in an in-office visit, including how to pick the best types of foods or ingredients for a given health condition, how to read and understand food labels, healthy recipes, how to track food and drink intake, and basic nutritional knowledge.
  Interventions: Behavioral: KP Personal Shopper Visits
- Office-Based Visit Arm (Active Comparator): 25 participants will be randomized to this arm. They will receive a baseline 30-minute phone call with the study dietitian to determine their current health problems, dietary patterns, shopping and cooking habits and health goals. They will then have 3 in-person visits with the dietitian conducted in an office at one of our medical office buildings. These in-person visits will be conducted monthly over a 3 month period. The information delivered in the visits will include how to pick the best types of foods or ingredients for a given health condition, how to read and understand food labels, healthy recipes, how to track food and drink intake, and basic nutritional knowledge.
  Interventions: Behavioral: In-Office Dietitian Visits

INTERVENTIONS:
Behavioral: KP Personal Shopper Visits — Testing co-shopping visits conducted in the grocery store (1:1 visits with dietitian while grocery shopping) versus in-office visits which are the current standard of care.
  Arms: Grocery-Store-Based Visit Arm
Behavioral: In-Office Dietitian Visits — Participants will have 3, 1 hour in-office sessions with the dietitian during which targeted curriculum on nutritional knowledge, weight management, healthier eating, menu and label reading, will be delivered. These visits will take place monthly over a three month period.
  Arms: Office-Based Visit Arm

SUMMARY:
Randomized trial of grocery-store based nutrition counseling visits for weight management vs. in-office visits. The investigators will test pre- and post-intervention individual-level dietary quality, knowledge, self-efficacy around dietary choice, and cost of shopping, measuring difference between intervention and control arms. At the study's end, the investigators will also conduct focus groups with a subset of 20 patients (10 from each arm) and do a structured interview with the dietitian to better understand the feasibility, strengths and shortcomings of this approach. Patients who complete the main portion of the trial will be randomly selected for recruitment into a focus group and consented separately for that focus group at the end of the study.

The investigators hypothesize that, compared to office-based visits, the KP Personal Shopper visits will result in higher member diet quality scores, better nutritional knowledge scores, higher self-efficacy and confidence around food purchasing decisions, and more favorable perception of the visit by both dietician and member. The KP Personal Shopper approach may also result in increased grocery store costs for some members. Long-term, the investigators hypothesize that improvements in member perception, knowledge and dietary quality will lead to improved health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Employee population of a specific Southeastern U.S. County
* 18-64 years of age
* Body Mass Index greater than or equal to 30kg/m^2 (Obese)
* Low rate of no-shows for office visits (<10%)
* Saw PCP or other provider in past 12 months
* Does at least 50% of the food shopping and/or food preparation for their household

Exclusion Criteria:

* non-English speaking
* Currently being treated for cancer (other than non-melanoma skin cancer)
* Pregnant or planning pregnancy in the next 6 months
* Had or considering having bariatric surgery
* Currently participating in commercial weight loss program (e.g. Jenny Craig)
* Currently enrolled in another weight management or nutrition study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Center for Health Research, Southeast, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Grocery-Store-Based Visit Arm: 28 participants were randomized to this arm. They were assigned to receive a baseline 30-minute phone call with the study dietitian to determine their current health problems, dietary patterns, shopping and cooking habits and health goals. They were then scheduled for 3 in-person visits with the dietitian conducted during grocery shopping trips at a local supermarket. These in-person visits were to be conducted monthly over a 3 month period. The information delivered in the visits was similar in content to that delivered in an in-office visit, including how to pick the best types of foods or ingredients for a given health condition, how to read and understand food labels, healthy recipes, how to track food and drink intake, and basic nutritional knowledge.
  KP Personal Shopper Visits: Testing co-shopping visits conducted in the grocery store (1:1 visits with dietitian while grocery shopping) versus in-office visits which are the current standard of care.
- Office-Based Visit Arm: 27 participants were randomized to this arm. They were assigned to receive a baseline 30-minute phone call with the study dietitian to determine their current health problems, dietary patterns, shopping and cooking habits and health goals. They were then scheduled for 3 in-person visits with the dietitian conducted at one of our medical office buildings. These in-person visits were conducted monthly over a 3 month period. The information delivered in the visits will included how to pick the best types of foods or ingredients for a given health condition, how to read and understand food labels, healthy recipes, how to track food and drink intake, and basic nutritional knowledge.
  In-Office Dietitian Visits: Participants will have 3, 1 hour in-office sessions with the dietitian during which targeted curriculum on nutritional knowledge, weight management, healthier eating, menu and label reading, will be delivered. These visits will take place monthly over a three month period.
Period: Overall Study
Arm/Group | Grocery-Store-Based Visit Arm | Office-Based Visit Arm
Started | 28 | 27
Completed | 25 | 25
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grocery-Store-Based Visit Arm | Office-Based Visit Arm | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10) | 43.4 (8.2) | 44.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 8 | 12 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 23 | 48
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 35.6 (4.7) | 34.1 (5.3) | 34.8 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dietary Quality Scores of Members as Measured Using the 2005 Healthy Eating Index (HEI).
Description: The Block FFQ will be administered at baseline in order to calculate a participant's baseline HEI score, and will be re-administered after the 3 month intervention to re-calculate the post-intervention HEI score.
  The numbers reported here represent the change from pre to post intervention, in the HEI scores for participants in each group
  HEI scores can range from 0 to 100, with 0 representing the least overall healthy diet, and 100 representing the most overall healthy diet. There are no units associated with the HEI score. The measure was developed by the US Dept of Agriculture and complete details regarding its development can be found on their website.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Grocery-Store-Based Visit Arm | Office-Based Visit Arm
Number analyzed (Participants) | 25 | 25
points | 5.2 (9.1) | 4.5 (9.7)

2. Secondary Outcome: Nutritional Knowledge of Members
Description: A modified version of the Parmenter-Wardle Nutrition Knowledge Questionnaire (1999, UK) has been created based on present-day guidelines and eating patterns in the Southeast U.S., and will be administered at baseline and scored, then re-administered after the intervention and re-scored to determine whether or how the score improved after the intervention with the dietitian.
Time Frame: 3 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Cost of Grocery Shopping for Members
Description: Receipts from a typical week's worth of grocery shopping will be collected from all participants at baseline. Then, the same process will be repeated each month during the intervention phase to see what effect participation has on costs of grocery shopping for participants (e.g. if buying more produce because shopping with dietitian - will shopping be more expensive?)
Time Frame: 3 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Member Self-efficacy and Confidence in Food Purchasing Decisions
Description: Will be assessed using a brief survey at baseline (scored) and re-surveyed after the intervention. Survey questions are based on similar items from other studies of health behavior interventions.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Grocery-Store-Based Visit Arm | Office-Based Visit Arm
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No